CLINICAL TRIAL: NCT07212166
Title: Psychometric and Linguistic Validation of PRO-AYA: Patient-Reported Outcomes for Adolescents and Young Adults (15-39) With Cancer
Brief Title: A Study of Questionnaires in Adolescents and Young Adults With Cancer
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 25-213
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Adolescents and Young Adults With Cancer
Keywords: PRO-AYA: Patient-Reported Outcomes for Adolescents and Young Adults; Psychometric and Linguistic Validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AYAs with cancer who are at least three months post treatment with no additional treatment planned: Complete via REDCap (at enrollment): PRO-AYA (PRO-AYA - Patient-Reported Outcomes for Adolescents and Young Adults), Patient-Reported ECOG PS, EORTC QLQ-C30, Demographic/Clinical Characteristics, Complete via REDCap (7-10 days later):
  PRO-AYA, Patient-Reported, ECOG PS
  Interventions: Other: Patient-Reported Outcome Surveys
- AYAs(Adolescents and Young Adults) who are fluent or prefer their healthcare be delivered in Spanish: Round 1 Cognitive Interviews Complete via REDCap: Spanish PRO-AYA, Demographic/Clinical Characteristic, Item modification based on patient feedback, Cohort 2b (n = 10) (AYAs who prefer healthcare delivery in Spanish) Round 2 Cognitive interviews, Complete via REDCap: Revised Spanish PRO-AYA, Demographic/Clinical Characteristics
  Interventions: Other: Spanish version of PRO-AYA and the cognitive interview

INTERVENTIONS:
Other: Patient-Reported Outcome Surveys — PRO-AYA , Patient-Reported ECOG PS, EORTC QLQ-C30, Demographic/Clinical Characteristics
  Groups: AYAs with cancer who are at least three months post treatment with no additional treatment planned
Other: Spanish version of PRO-AYA and the cognitive interview — Revised Spanish PRO-AYA, Demographic/Clinical Characteristics
  Groups: AYAs(Adolescents and Young Adults) who are fluent or prefer their healthcare be delivered in Spanish

SUMMARY:
The purpose of this study is to evaluate a questionnaire called PRO-AYA: Patient-Reported Outcomes for Adolescents and Young Adults.

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish proficient

  o As assessed by two items: How well do you speak English? What is your preferred language for healthcare?
* Diagnosed with the first instance of a cancer or the relapse of a prior cancer between the ages of 15 - 39
* Able to complete questionnaires by themselves or with assistance
* ECOG Performance Status (0-4)
* 3 months from last treatment without plan to initiate any form of cancer-directed treatment in the next 3 months

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at MSK.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Test-retest reliability | up to one month
  The test-retest reliability will be based on the intraclass correlation (ICC) coefficients between the baseline and follow-up domain scores of PRO-AYA.
Linguistically validate PRO-AYA or patients who prefer their healthcare be delivered in Spanish. (Cohort 2) | up to a month
  The primary goal of these cognitive interviews is to ensure that the wording and/or phrasing of the instructions, questions and answer choices are appropriate for native Spanish-speakers. The wording and phrasing are a result of direct translation of the English version of the PRO-AYA to a Spanish version.

CONTACTS AND LOCATIONS:
Overall Officials: Viswatej Avutu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm